CLINICAL TRIAL: NCT02061293
Title: A Double-Blind Trial of Psilocybin-Assisted Treatment of Alcohol Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Heffter Research Institute (Other); University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-00614; Heffter 113080-2 (Other Grant/Funding Number: Heffter Research Institute)
Record Dates: First submitted 2014-02-07; First posted 2014-02-12 (Estimated); Results first posted 2022-10-18 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Alcohol Dependence
MeSH Terms: conditions — Alcoholism | interventions — Psilocybin; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Psilocybin (Experimental): Psilocybin 25 mg/70 kg PO administered at week 4, 25-40 mg/70 kg PO administered at week 8.
  Interventions: Drug: Psilocybin; Behavioral: Motivational Enhancement and Taking Action (META)
- Diphenhydramine (Active Comparator): Diphenhydramine 50 mg PO administered at week 4, 50-100 mg PO administered at week 8.
  Interventions: Drug: Diphenhydramine; Behavioral: Motivational Enhancement and Taking Action (META)

INTERVENTIONS:
Drug: Psilocybin
  Arms: Psilocybin
Drug: Diphenhydramine
  Arms: Diphenhydramine
Behavioral: Motivational Enhancement and Taking Action (META) — Manualized psychosocial intervention based on motivational enhancement therapy, functional analysis, and implementation of a change plan.

SUMMARY:
Several lines of evidence suggest that classic hallucinogens such as psilocybin can facilitate behavior change in addictions such as alcohol dependence. The proposed investigation is a multi-site, double-blind active-controlled trial (n = 180, 90 per group) contrasting the acute and persisting effects of psilocybin to those of diphenhydramine in the context of outpatient alcoholism treatment.

DETAILED DESCRIPTION:
Two to four sites will participate in this study. Aims of the study are 1) to characterize the acute effects of PO psilocybin 25 mg/70 kg, 30 mg/70 kg, and 40 mg/70 kg in alcohol dependent patients; 2) to evaluate the effect of psilocybin treatment on drinking outcomes for 32 weeks after the first administration, relative to diphenhydramine control; 3) to test whether or not characteristics of the drug administration session experiences mediate effects of psilocybin on short-term (1 week) persisting effects and post-session drinking behavior, 4) to evaluate the explanatory value of changes in alcohol craving, self-efficacy, motivation, and other psychological domains in accounting for the observed experimental effect of psilocybin relative to diphenhydramine control, and 5) to evaluate pre-post changes in drinking in participants after they receive psilocybin in the third session.

The total duration of psychosocial treatment in the double-blind period will be 12 weeks, and double-blind drug administration sessions will occur after 4 and 8 weeks. In the first psilocybin session, a dose of 25 mg/70 kg will be administered. Depending on the response in the first session, the dose for the second session may be increased to 30 mg/70 kg or 40 mg/70 kg, or held at 25mg/70kg. The dose of diphenhydramine will start at 50 mg, and may be increased to 100 mg or held at 50 mg in the second session, depending on response in the first session. Following completion of the double-blind period (34 weeks after randomization) all participants who meet interim safety criteria will be offered an additional session in which psilocybin will be administered. The drug will be administered during 8-hour sessions in an outpatient setting under close medical and psychiatric monitoring. The drug administration sessions will occur in the context of an extended version of Motivational Enhancement Therapy (Motivational Enhancement and Taking Action, META) with the addition of standardized preparation before and debriefing and follow-up after the psilocybin administration sessions. Extensive screening and baseline assessment will be completed, including thorough safety screening and assessment of participant characteristics that could potentially moderate treatment response. Within-session and short-term persisting effects will be assessed. Drinking outcomes and changes in several potential mediators of treatment effect, including motivation, self-efficacy, craving, depression, anxiety, and spiritual dimensions of the experience, will be measured until 50 weeks after the first drug administration session, for a total of 54 weeks from the initiation of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females age 25-65 with SCID (DSM-IV) diagnosis of alcohol dependence who
2. Want to stop or decrease their drinking
3. Are not participating in any formal treatment for alcohol dependence (12-step meetings are not considered treatment)
4. Are able to provide voluntary informed consent
5. Have at least 4 heavy drinking days in the past 30 days
6. If female of childbearing potential, are willing to use approved form of contraception from screening until after the psilocybin administration sessions
7. Have a family member or friend who can pick them up and stay with them overnight after the psilocybin administration sessions
8. Are able to provide adequate locator information.

Exclusion Criteria:

1. Medical conditions that would preclude safe participation in the trial (e.g., seizure disorder, significantly impaired liver function, coronary artery disease, heart failure, uncontrolled hypertension (above 165/95 mmHg at screening), history of cerebrovascular accident, asthma, hyperthyroidism, narrow-angle glaucoma, stenosing peptic ulcer, pyloroduodenal obstruction, symptomatic prostatic hypertrophy, or bladder-neck obstruction)
2. Exclusionary psychiatric conditions (schizophrenia, schizoaffective disorder, bipolar disorder, current major depressive episode, current post-traumatic stress disorder, current suicidality or history of medically serious suicide attempt)
3. Cognitive impairment (Folstein Mini Mental State Exam score < 26)
4. A family history of schizophrenia or schizoaffective disorder (first or second degree relatives), or bipolar disorder type 1 (first degree relatives)
5. History of hallucinogen use disorder, or any use in the past 1 year, or >25 lifetime uses;
6. Cocaine, psychostimulant, opioid, or cannabis dependence (past 12 months)
7. Current non-medical use of cocaine, psychostimulants, or opioids (past 30 days)
8. Significant alcohol withdrawal (CIWA-Ar score greater than 7. Patients presenting at screening in withdrawal may be referred for detoxification and reassessed within 30 days)
9. Serious ECG abnormalities (e.g., evidence of ischemia, myocardial infarction, QTc prolongation [QTc > .045 for men, QTc > .047 for women])
10. Serious abnormalities of complete blood count or chemistries
11. Active legal problems with the potential to result in incarceration
12. Pregnancy or lactation
13. Need to take medication with significant potential to interact with study medications (e.g., antidepressants, antipsychotics, psychostimulants, treatments for addictions, other dopaminergic or serotonergic agents, lithium, anticonvulsants).
14. Allergy or hypersensitivity to psilocybin or diphenhydramine.
15. High risk of adverse emotional or behavioral reaction based on investigator's clinical evaluation (e.g., evidence of serious personality disorder, antisocial behavior, serious current stressors, lack of meaningful social support).

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Bogenschutz, MD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - Clinical and Translational Science Institute, NYU Langone Medical Center, New York, New York

REFERENCES:
- [Derived] Pagni BA, Petridis PD, Podrebarac SK, Grinband J, Claus ED, Bogenschutz MP. Psilocybin-induced changes in neural reactivity to alcohol and emotional cues in patients with alcohol use disorder: an fMRI pilot study. Sci Rep. 2024 Feb 7;14(1):3159. doi: 10.1038/s41598-024-52967-8. PMID 38326432
- [Derived] Agin-Liebes G, Nielson EM, Zingman M, Kim K, Haas A, Owens LT, Rogers U, Bogenschutz M. Reports of self-compassion and affect regulation in psilocybin-assisted therapy for alcohol use disorder: An interpretive phenomenological analysis. Psychol Addict Behav. 2024 Feb;38(1):101-113. doi: 10.1037/adb0000935. Epub 2023 Jun 5. PMID 37276086
- [Derived] O'Donnell KC, Mennenga SE, Owens LT, Podrebarac SK, Baron T, Rotrosen J, Ross S, Forcehimes AA, Bogenschutz MP. Psilocybin for alcohol use disorder: Rationale and design considerations for a randomized controlled trial. Contemp Clin Trials. 2022 Dec;123:106976. doi: 10.1016/j.cct.2022.106976. Epub 2022 Nov 2. PMID 36332827
- [Derived] Bogenschutz MP, Ross S, Bhatt S, Baron T, Forcehimes AA, Laska E, Mennenga SE, O'Donnell K, Owens LT, Podrebarac S, Rotrosen J, Tonigan JS, Worth L. Percentage of Heavy Drinking Days Following Psilocybin-Assisted Psychotherapy vs Placebo in the Treatment of Adult Patients With Alcohol Use Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2022 Oct 1;79(10):953-962. doi: 10.1001/jamapsychiatry.2022.2096. PMID 36001306
- [Derived] Bogenschutz MP, Forcehimes AA, Pommy JA, Wilcox CE, Barbosa PC, Strassman RJ. Psilocybin-assisted treatment for alcohol dependence: a proof-of-concept study. J Psychopharmacol. 2015 Mar;29(3):289-99. doi: 10.1177/0269881114565144. Epub 2015 Jan 13. PMID 25586396

RESULTS

PARTICIPANT FLOW:
Groups:
- Psilocybin: Psilocybin 25 mg/70 kg PO administered at week 4, 25-40 mg/70 kg PO administered at week 8.
  Psilocybin
  Motivational Enhancement and Taking Action (META): Manualized psychosocial intervention based on motivational enhancement therapy, functional analysis, and implementation of a change plan.
- Diphenhydramine: Diphenhydramine 50 mg PO administered at week 4, 50-100 mg PO administered at week 8.
  Diphenhydramine
  Motivational Enhancement and Taking Action (META): Manualized psychosocial intervention based on motivational enhancement therapy, functional analysis, and implementation of a change plan.
Period: Overall Study
Arm/Group | Psilocybin | Diphenhydramine
Started | 49 | 46
Completed | 48 | 45
Not Completed | 1 | 1
Not completed — Elevated Blood Pressure | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Psilocybin | Diphenhydramine | Total
Number analyzed (Participants) | 48 | 45 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.94 (10.91) | 44.24 (12.15) | 45.59 (11.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 28 | 24 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 8 | 14
  Not Hispanic or Latino | 42 | 37 | 79
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 37 | 36 | 73
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 7 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 48 | 45 | 93

OUTCOME MEASURES:

1. Primary Outcome: Percent of Heavy Drinking Days
Description: The Timeline Follow-back (TLFB) method is used to calculate the percent of heavy drinking days. The TLFB is a method for assessing the number of drinks of alcohol on a daily basis over the previous 30 days. For each day in the recall period, the participant indicates the number of drinks of alcohol they consumed. The TLFB provides a calendar prompt and number of other memory aids (e.g., holidays, payday, and other personally relevant dates) to facilitate accurate recall of drug use during the target period. Heavy drinking is defined as ≥4 drinks per day for women and ≥5 drinks per day for men.
Time Frame: Screening (Week 0)
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Psilocybin | Diphenhydramine
Number analyzed (Participants) | 48 | 45
percentage of days | 56.48 (31.77) | 48.57 (28.73)

2. Primary Outcome: Percent of Heavy Drinking Days
Description: as for outcome 1
Time Frame: Baseline (Week 4)
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Psilocybin | Diphenhydramine
Number analyzed (Participants) | 48 | 45
percentage of days | 24.11 (26.29) | 21.31 (20.14)

3. Primary Outcome: Percent of Heavy Drinking Days
Description: as for outcome 1
Time Frame: Follow Up (Weeks 5-36)
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Psilocybin | Diphenhydramine
Number analyzed (Participants) | 48 | 45
percentage of days | 9.71 (26.21) | 23.57 (26.67)

4. Primary Outcome: Drinks Per Day
Description: The Timeline Follow-back (TLFB) method is used to calculate drinks per day. The TLFB is a method for assessing the number of drinks of alcohol on a daily basis over the previous 30 days. For each day in the recall period, the participant indicates the number of drinks of alcohol they consumed. The TLFB provides a calendar prompt and number of other memory aids (e.g., holidays, payday, and other personally relevant dates) to facilitate accurate recall of drug use during the target period.
Time Frame: Screening (Week 0)
Measure: Mean (Standard Deviation); unit: drinks per day
Arm/Group | Psilocybin | Diphenhydramine
Number analyzed (Participants) | 48 | 45
drinks per day | 5.2 (2.81) | 4.38 (2.39)

5. Primary Outcome: Drinks Per Day
Description: as for outcome 4
Time Frame: Baseline (Week 4)
Measure: Mean (Standard Deviation); unit: drinks per day
Arm/Group | Psilocybin | Diphenhydramine
Number analyzed (Participants) | 48 | 45
drinks per day | 2.77 (2.3) | 2.19 (1.98)

6. Primary Outcome: Drinks Per Day
Description: as for outcome 4
Time Frame: Follow Up (Weeks 5-36)
Measure: Mean (Standard Deviation); unit: drinks per day
Arm/Group | Psilocybin | Diphenhydramine
Number analyzed (Participants) | 48 | 45
drinks per day | 1.17 (1.99) | 2.26 (2.02)

7. Primary Outcome: Percent of Drinking Days
Description: The Timeline Follow-back (TLFB) method is used to calculate the percentage of days that participants drank alcohol. The TLFB is a method for assessing the number of drinks of alcohol on a daily basis over the previous 30 days. For each day in the recall period, the participant indicates the number of drinks of alcohol they consumed. The TLFB provides a calendar prompt and number of other memory aids (e.g., holidays, payday, and other personally relevant dates) to facilitate accurate recall of drug use during the target period.
Time Frame: Screening (Week 0)
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Psilocybin | Diphenhydramine
Number analyzed (Participants) | 48 | 45
percentage of days | 78.03 (27.02) | 71.68 (28.98)

8. Primary Outcome: Percent of Drinking Days
Description: as for outcome 7
Time Frame: Baseline (Week 4)
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Psilocybin | Diphenhydramine
Number analyzed (Participants) | 48 | 45
percentage of days | 52.98 (31.78) | 45.99 (30.4)

9. Primary Outcome: Percent of Drinking Days
Description: as for outcome 7
Time Frame: Follow Up (Weeks 5-36)
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Psilocybin | Diphenhydramine
Number analyzed (Participants) | 48 | 45
percentage of days | 29.39 (32.86) | 42.83 (33.43)

10. Secondary Outcome: Short Inventory of Problems (SIP-2R) Score
Description: 15-item self-report questionnaire assessing problems related to alcohol use. Items are ranked on a 4-point Likert scale ranging from 0 (never) to 3 (daily or almost daily). The total score range is 0-45; the higher the score, the more problems related to alcohol use.
Time Frame: Baseline (Week 4)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psilocybin | Diphenhydramine
Number analyzed (Participants) | 47 | 45
score on a scale | 20.26 (8.89) | 21.6 (9.61)

11. Secondary Outcome: Short Inventory of Problems (SIP-2R) Score
Description: as for outcome 10
Time Frame: Week 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psilocybin | Diphenhydramine
Number analyzed (Participants) | 44 | 40
score on a scale | 6.59 (8.8) | 13 (10.48)

12. Secondary Outcome: Percentage of Participants Achieving Abstinence From Drinking
Description: The Timeline Follow-back (TLFB) method is used in calculating abstinence from drinking. The TLFB is a method for assessing the number of drinks of alcohol on a daily basis over the previous 30 days. For each day in the recall period, the participant indicates the number of drinks of alcohol they consumed. The TLFB provides a calendar prompt and number of other memory aids (e.g., holidays, payday, and other personally relevant dates) to facilitate accurate recall of drug use during the target period. Abstinence is defined as zero drinks of alcohol over the target period.
Time Frame: From Week 5 (1 week after first drug administration) up to Week 36
Measure: Number; unit: Percentage of participants
Arm/Group | Psilocybin | Diphenhydramine
Number analyzed (Participants) | 48 | 45
Percentage of participants | 22.9 | 8.9

13. Secondary Outcome: Percentage of Participants Achieving Abstinence From Drinking
Description: as for outcome 12
Time Frame: From Week 33 up to Week 36
Measure: Number; unit: Percentage of participants
Arm/Group | Psilocybin | Diphenhydramine
Number analyzed (Participants) | 48 | 45
Percentage of participants | 47.9 | 24.4

14. Secondary Outcome: Percent of Participants Achieving No Heavy Drinking Days
Description: The Timeline Follow-back (TLFB) method is used in calculating the number of heavy drinking days. The TLFB is a method for assessing the number of drinks of alcohol on a daily basis over the previous 30 days. For each day in the recall period, the participant indicates the number of drinks of alcohol they consumed. The TLFB provides a calendar prompt and number of other memory aids (e.g., holidays, payday, and other personally relevant dates) to facilitate accurate recall of drug use during the target period. Heavy drinking is defined as ≥4 drinks per day for women and ≥5 drinks per day for men.
Time Frame: From Week 5 (1 week after first drug administration) up to Week 36
Measure: Number; unit: Percentage of participants
Arm/Group | Psilocybin | Diphenhydramine
Number analyzed (Participants) | 48 | 45
Percentage of participants | 33.3 | 11.1

15. Secondary Outcome: Percent of Participants Achieving No Heavy Drinking Days
Description: as for outcome 14
Time Frame: From Week 33 Up to Week 36
Measure: Number; unit: Percentage of participants
Arm/Group | Psilocybin | Diphenhydramine
Number analyzed (Participants) | 48 | 45
Percentage of participants | 62.5 | 40

16. Secondary Outcome: Percent of Participants Achieving WHO Risk Drinking Level Decrease of at Least 1 Level
Description: For men, WHO low risk drinking (level 1) is defined as >0 grams of alcohol/day (g/d) to 40 g/d; moderate risk (level 2) as >40 g/d to 60 g/d; high risk (level 3) as >60 g/d to 100 g/d; and very high risk (level 4) as >100 g/d. For women, low risk (level 1) is defined as >0 g/d to 20 g/d; moderate risk (level 2) as >20 g/d to 40 g/d; high risk (level 3) as >40 g/d to 60 g/d; and very high risk (level 4) as >60 g/d. Abstinence was defined as no risk (level 0).
Time Frame: From Week 5 (1 week after first drug administration) up to Week 36
Measure: Number; unit: Percentage of participants
Arm/Group | Psilocybin | Diphenhydramine
Number analyzed (Participants) | 48 | 45
Percentage of participants | 83.3 | 71.1

17. Secondary Outcome: Percent of Participants Achieving WHO Risk Drinking Level Decrease of at Least 1 Level
Description: as for outcome 16
Time Frame: From Week 33 Up to Week 36
Measure: Number; unit: Percentage of participants
Arm/Group | Psilocybin | Diphenhydramine
Number analyzed (Participants) | 48 | 45
Percentage of participants | 89.6 | 64.4

18. Secondary Outcome: Percent of Participants Achieving WHO Risk Drinking Level Decrease of at Least 2 Levels
Description: as for outcome 16
Time Frame: From Week 5 (1 week after first drug administration) up to Week 36
Measure: Number; unit: Percentage of participants
Arm/Group | Psilocybin | Diphenhydramine
Number analyzed (Participants) | 48 | 45
Percentage of participants | 60.4 | 40

19. Secondary Outcome: Percent of Participants Achieving WHO Risk Drinking Level Decrease of at Least 2 Levels
Description: as for outcome 16
Time Frame: From Week 33 Up to Week 36
Measure: Number; unit: Percentage of participants
Arm/Group | Psilocybin | Diphenhydramine
Number analyzed (Participants) | 48 | 45
Percentage of participants | 60.4 | 40

20. Secondary Outcome: Percent of Participants Achieving WHO Risk Drinking Level Decrease of at Least 3 Levels
Description: as for outcome 16
Time Frame: From Week 5 (1 week after first drug administration) up to Week 36
Measure: Number; unit: Percentage of participants
Arm/Group | Psilocybin | Diphenhydramine
Number analyzed (Participants) | 48 | 45
Percentage of participants | 29.92 | 13.3

21. Secondary Outcome: Percent of Participants Achieving WHO Risk Drinking Level Decrease of at Least 3 Levels
Description: as for outcome 16
Time Frame: From Week 33 up to Week 36
Measure: Number; unit: Percentage of participants
Arm/Group | Psilocybin | Diphenhydramine
Number analyzed (Participants) | 48 | 45
Percentage of participants | 37.5 | 17.8

ADVERSE EVENTS:
Time Frame: After first medication administration (week 4) through week 36.
Description: Study team / PI monitor AEs at every assessment visit.
Arm/Group | Psilocybin | Diphenhydramine
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/48 | 2/45
Other Adverse Events (participants affected / at risk) | 37/48 | 29/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Psilocybin (N=48) | Diphenhydramine (N=45)
Mallory-Weiss Syndrom (Gastrointestinal disorders) | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Psilocybin (N=48) | Diphenhydramine (N=45)
Anemia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Photopsia (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 2
Diverticulitis (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 10 | 4
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1
Asthenia (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Influenza like Illness (General disorders) | 0 | 1
Oedema (General disorders) | 0 | 1
Pain (General disorders) | 1 | 3
Peripheral swelling (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Dermatitis contact (Immune system disorders) | 0 | 1
Food allergy (Immune system disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 3
Bronchitis bacterial (Infections and infestations) | 0 | 1
Corona virus infection (Infections and infestations) | 2 | 0
Eye infection (Infections and infestations) | 0 | 1
Fungal infection (Infections and infestations) | 0 | 1
Gingivitis (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 1 | 2
Pneumonia (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Viral upper resp. tract infection (Infections and infestations) | 2 | 3
Alcohol poisoning (Injury, poisoning and procedural complications) | 2 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Traumatic lung injury (Injury, poisoning and procedural complications) | 0 | 1
Biopsy cervix (Investigations) | 1 | 0
Blood pressure diastolic increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 21 | 2
Hypoesthesia (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0
Sedation (Nervous system disorders) | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 2
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 2
Anger (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 7 | 1
Depressed mood (Psychiatric disorders) | 3 | 2
Depression (Psychiatric disorders) | 2 | 2
Dysphoria (Psychiatric disorders) | 1 | 0
Illusion (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 3 | 2
Restlessness (Psychiatric disorders) | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 4 | 2
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Testicular pain (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lower resp. tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sexual abuse (Social circumstances) | 0 | 1
Arthoscopic surgery (Surgical and medical procedures) | 0 | 1
Endodontic procedure (Surgical and medical procedures) | 0 | 1
Skin cosmetic procedure (Surgical and medical procedures) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/93/NCT02061293/Prot_SAP_000.pdf